CLINICAL TRIAL: NCT06767709
Title: AID-OMIE - Artificial Intelligence in Detection of Occlusive Myocardial Infarction in Emergency Medicine
Acronym: AID-OMIE
Status: Not yet recruiting | Type: Observational
Sponsor: Institute of Mountain Emergency Medicine (Other)
Responsible Party: Principal Investigator, Simon Rauch, Senior Researcher, Institute of Mountain Emergency Medicine
Other Study IDs: 01-2025
Record Dates: First submitted 2025-01-05; First posted 2025-01-10 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Cardiac Arrest, Out-Of-Hospital; Cardiac Arrest Due to Underlying Cardiac Condition
Keywords: Cardiac arrest; OHCA; Occlusion myocardial infarction; OMI; Artificial intelligence
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients after Out-of-Hospital Cardiac Arrest (OHCA) with ROSC in the Province of Bolzano, Italy: Patients after Out-of-Hospital Cardiac Arrest (OHCA) with Return of Spontaneous Circulation (ROSC) in the Province of Bolzano, Italy

SUMMARY:
Study Objective and Hypothesis The study hypothesizes that artificial intelligence (AI)-assisted interpretation of the 12-lead electrocardiogram (ECG) can improve the care of patients resuscitated after out-of-hospital cardiac arrest (OHCA) by enabling faster and more accurate detection of occlusion myocardial infarction (OMI). This enhanced diagnostic approach could reduce the time required for revascularization, improve patient outcomes, and decrease unnecessary activations of cardiac catheterization laboratories. The primary objective of the study is to assess the effectiveness of an AI-powered ECG model in identifying acute OMI in OHCA patients whose post-return of spontaneous circulation (ROSC) ECG does not show ST-elevation.

Methods

This is a retrospective observational study involving OHCA patients in Bolzano, Italy, who meet the following inclusion criteria:

Aged 18 years or older. Achieved ROSC after cardiac arrest. Underwent coronary angiography (CAG) within seven days post-OHCA. Prehospital post-ROSC ECG and CAG reports available.

Exclusion criteria include in-hospital cardiac arrest (IHCA), traumatic cardiac arrest, cardiac arrest from a non-cardiac cause, and poor-quality or corrupted ECG images. Post-ROSC ECGs will be analyzed using the PMcardio App, an AI tool for ECG interpretation. The data will be fully anonymized before storage. Coronary angiography charts will be reviewed for the presence of atherosclerotic lesions, the degree of arterial narrowing, and Thrombolysis in Myocardial Infarction (TIMI) flow, which assesses blood flow in coronary arteries.

Study Outcomes The primary outcome is the sensitivity and specificity of the AI-assisted ECG in detecting OMI in patients whose post-ROSC ECG does not show ST-elevation. Secondary outcomes include the frequency of OMI in OHCA patients without ST-elevation and the ability of the AI model to rule out OMI accurately in these cases.

DETAILED DESCRIPTION:
Study Objective and Hypothesis The study hypothesizes that artificial intelligence (AI)-assisted interpretation of the 12-lead electrocardiogram (ECG) can improve the care of patients resuscitated after out-of-hospital cardiac arrest (OHCA) by enabling faster and more accurate detection of occlusion myocardial infarction (OMI). This enhanced diagnostic approach could reduce the time required for revascularization, improve patient outcomes, and decrease unnecessary activations of cardiac catheterization laboratories. The primary objective of the study is to assess the effectiveness of an AI-powered ECG model in identifying acute OMI in OHCA patients whose post-return of spontaneous circulation (ROSC) ECG does not show ST-elevation.

Methods

This is a retrospective observational study involving OHCA patients in Bolzano, Italy, who meet the following inclusion criteria:

OHCA from 2018-2025 Aged 18 years or older. Achieved ROSC after cardiac arrest. Underwent coronary angiography (CAG) within seven days post-OHCA. Prehospital post-ROSC ECG and CAG reports available.

Exclusion criteria include in-hospital cardiac arrest (IHCA), traumatic cardiac arrest, cardiac arrest from a non-cardiac cause, and poor-quality or corrupted ECG images. Post-ROSC ECGs will be analyzed using the PMcardio App, an AI tool for ECG interpretation. The data will be fully anonymized before storage. Coronary angiography charts will be reviewed for the presence of atherosclerotic lesions, the degree of arterial narrowing, and Thrombolysis in Myocardial Infarction (TIMI) flow, which assesses blood flow in coronary arteries.

Study Outcomes The primary outcome is the sensitivity and specificity of the AI-assisted ECG in detecting OMI in patients whose post-ROSC ECG does not show ST-elevation. Secondary outcomes include the frequency of OMI in OHCA patients without ST-elevation and the ability of the AI model to rule out OMI accurately in these cases.

ELIGIBILITY:
Inclusion Criteria:

* OHCA from with ROSC in the Province of Bolzano, Italy
* Coronary angiography (CAG) within 7 days post-OHCA
* Age > 18 years
* Available prehospital post-ROSC ECG
* Available CAG report

Exclusion Criteria:

* In-Hospital Cardiac Arrest (IHCA)
* Age < 18 years
* Traumatic cardiac arrest
* Cardiac arrest from a clear non-cardiac cause
* Corrupted ECG images
* Poor ECG digitalization quality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who suffered OHCA from presumed cardiac cause and sustained ROSC.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of detecting OMI from the post-ROSC ECG with AI-assisted ECG interpretation in patients following OHCA with ROSC, where the post-ROSC ECG does not show ST-elevation. | Within 7 days after OHCA
  Sensitivity and specificity of detecting occlusion myocardial infarction (OMI) from the electrocardiogram (ECG) taken after return of spontaneous circulation (ROSC) using artificial intelligence (AI)-assisted ECG interpretation in patients resuscitated from out-of-hospital cardiac arrest (OHCA) with ROSC, where the post-ROSC ECG does not display ST-segment elevation.

SECONDARY OUTCOMES:
Frequency of OMI post-OHCA without ST-elevation in the post-ROSC ECG | Within 7 days after OHCA
  Frequency of occlusion myocardial infarction (OMI) in patients resuscitated from out-of-hospital cardiac arrest (OHCA) who achieved return of spontaneous circulation (ROSC), where the electrocardiogram (ECG) recorded post-ROSC does not show ST-segment elevation.
Sensitivity and specificity of excluding OMI with AI-assisted ECG interpretation in patients following OHCA with ROSC, where the post-ROSC ECG does not show ST-elevation. | Within 7 days from OHCA
  Sensitivity and specificity of ruling out occlusion myocardial infarction (OMI) using artificial intelligence (AI)-assisted electrocardiogram (ECG) interpretation in patients resuscitated from out-of-hospital cardiac arrest (OHCA) who achieved return of spontaneous circulation (ROSC), where the post-ROSC ECG does not display ST-segment elevation.

IPD SHARING:
Plan to Share IPD: No